CLINICAL TRIAL: NCT02112331
Title: Influence of Physical Treatments of Human Milk on the Kinetics of Gastric Lipolysis in Preterm Newborns
Acronym: ARCHILACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2013-A01460-45
Record Dates: First submitted 2014-03-25; First posted 2014-04-11 (Estimated); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Premature Birth
Keywords: Preterm newborns; Gastric lipolysis; Physical treatments; Human milk
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Raw human milk / pasteurized human milk (Experimental): Raw human milk compared to pasteurized human milk. Two meals administration (20mL/kg) per day during 6 days in a randomized order, with an intragastric tube : one with raw milk and one with pasteurized milk.
  In order to characterise gastric effluents at different postprandial times after ingestion and to measure gastric lipolysis and proteolysis, at each administration two gastric samples will be collected with the intragastric tube :
  * one before the meal,
  * and one either 35, 60 or 90 minutes (randomized time frame) after the meal.
  Interventions: Other: Raw human milk; Other: Pasteurized human milk; Other: Gastric samples
- Pasteurized human milk / pasteurized-homogenized human milk (Experimental): Pasteurized human milk compared to pasteurized-homogenized human milk. Two meals administration (20mL/kg) per day during 6 days in a randomized order, with an intragastric tube : one with pasteurized milk and one with pasteurized-homogenized milk.
  In order to characterise gastric effluents at different postprandial times after ingestion and to measure gastric lipolysis and proteolysis, at each administration two gastric samples will be collected with the intragastric tube :
  * one before the meal,
  * and one either 35, 60 or 90 minutes (randomized time frame) after the meal.
  Interventions: Other: Pasteurized human milk; Other: Pasteurized-homogenized human milk; Other: Gastric samples

INTERVENTIONS:
Other: Raw human milk
  Arms: Raw human milk / pasteurized human milk
Other: Pasteurized human milk
Other: Pasteurized-homogenized human milk
  Arms: Pasteurized human milk / pasteurized-homogenized human milk
Other: Gastric samples

SUMMARY:
The optimization of newborns nutrition is a challenge especially for preterm newborns for whom nutrition plays a crucial part in cerebral and global development. Human milk is considered as the best food for newborns. Several short and long-term beneficial health effects were attributed to breastfeeding and have induced the increase of human milk in preterm newborns nutrition.

Whereas the chemical composition of infant formula has been optimized to mimic human milk, there is still a major difference between the structure of human milk and commercial infant formulas. It is well known in adult nutrition that the structure of emulsions influences their susceptibility to hydrolysis, such results have been obtained either on in vitro or in vivo studies.

Human milk is a natural emulsion (oil in water). Lipids droplets are dispersed under the form of entities called milk fat globules (average diameter 4 µm, span 0.1-20 μm). The globules are stabilized by a trilayered membrane composed mainly of polar lipids (phospholipids, sphingolipids and gangliosides), of proteins, neutral lipids and other minor compounds.

The physical treatments apply to human milk or more generally to bovine milk to pasteurize or stabilize the milk modify the structure of the natural emulsion. Heat treatment for instance induces whey proteins denaturation and the adsorption of protein aggregates on the surface of the milk fat globules. Heat treatment also leads to the denaturation of bile salt stimulated lipase. These effects limit intragastric lipolysis in preterm newborns.

Conversely, reduction of milk globules size, by homogenisation of milk, increases the specific surface available for lipase adsorption and limits the lost of fat during enteral administration of milk. Such treatment could thus enhance gastric lipolysis and improve fat absorption of preterm newborns.

The objective of this trial is to evaluate the effects of physical treatments (pasteurization and homogenisation by ultrasonication) applied to human milk on gastric lipolysis and milk destructuration. This trial is conducted, in vivo, on preterm newborns.

ELIGIBILITY:
Inclusion Criteria:

* Premature neonates born before 32 weeks of gestation
* Newborn dwelled near Rennes
* Volume of enteral nutrition > 120 mL/kg/j (Day 0)
* Written-informed parental consent for the study

Exclusion Criteria:

* Digestive congenital anomalies
* Antecedent of enterocolitis
* Patient included in other study
* Abdominal distension on Day 0
* Treatment by morphine or catecholamine on Day 0

Ages: 5 Days to 21 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2014-04; Primary Completion 2015-08 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Percentage of triacylglycerol hydrolysis | 35 min
  Monitoring of the lipolysis kinetics, using chromatography methods

SECONDARY OUTCOMES:
Size distribution and specific surface of milk fat globule by laser light scattering | 35 min, 60 min, 90 min
Fat composition | 35 min, 60 min, 90 min
  Fat composition by chromatographic techniques : High-Performance Liquid Chromatography (HPLC), Gas Chromatography (GC)
Lipolysis products | 35 min, 60 min, 90 min
  Lipolysis products by thin layer chromatography (TLC), gas chromatography (GC) and IATROSCAN
Proteolysis products | 35 min, 60 min, 90 min
  Proteolysis products by electrophoresis (SDS-Page) and free amino acids by chromatography (HPLC)
Kinetic of the gastric emptying | 35 min, 60 min, 90 min
  Evaluation of the kinetic of the gastric emptying by measuring the volume remaining in the stomach
Lipolysis level | 35 min, 60 min, 90 min
  Comparison of lipolysis level obtained either on in vitro or in vivo studies
Percentage of triacylglycerol hydrolysis | 60 min, 90 min
Percentage of free fatty acids appearing | 35 min, 60 min, 90 min
  Monitoring of the lipolysis kinetics, using chromatography methods

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Pladys, MD, PhD, Principal Investigator — Pôle de pédiatrie, CHU de Rennes, FRANCE; Didier Dupont, Study Chair — Agrocampus Ouest - Département AgroAlimentaire UMR 1253 INRA " Science et Technologie du Lait et de l'Oeuf ", Rennes, FRANCE
Locations (1):
- Rennes University Hospital, Rennes, France

REFERENCES:
- [Background] de Oliveira SC, Bourlieu C, Menard O, Bellanger A, Henry G, Rousseau F, Dirson E, Carriere F, Dupont D, Deglaire A. Impact of pasteurization of human milk on preterm newborn in vitro digestion: Gastrointestinal disintegration, lipolysis and proteolysis. Food Chem. 2016 Nov 15;211:171-9. doi: 10.1016/j.foodchem.2016.05.028. Epub 2016 May 6. PMID 27283620
- [Derived] de Oliveira SC, Bellanger A, Menard O, Pladys P, Le Gouar Y, Henry G, Dirson E, Rousseau F, Carriere F, Dupont D, Bourlieu C, Deglaire A. Impact of homogenization of pasteurized human milk on gastric digestion in the preterm infant: A randomized controlled trial. Clin Nutr ESPEN. 2017 Aug;20:1-11. doi: 10.1016/j.clnesp.2017.05.001. Epub 2017 May 15. PMID 29072162
- [Derived] de Oliveira SC, Bellanger A, Menard O, Pladys P, Le Gouar Y, Dirson E, Kroell F, Dupont D, Deglaire A, Bourlieu C. Impact of human milk pasteurization on gastric digestion in preterm infants: a randomized controlled trial. Am J Clin Nutr. 2017 Feb;105(2):379-390. doi: 10.3945/ajcn.116.142539. Epub 2017 Jan 4. PMID 28052887